CLINICAL TRIAL: NCT03463954
Title: Prospective, Multicenter Confirmatory Clinical Evaluation of Novilase® Interstitial Laser Therapy for the Focal Destruction of Malignant Breast Tumors ≤15 mm (BR-003)
Brief Title: Confirmatory Clinical Evaluation of Novilase® Laser Therapy for Focal Destruction of Malignant Breast Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novian Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-003
Record Dates: First submitted 2018-01-23; First posted 2018-03-13 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Malignant Neoplasm of Breast
Keywords: less than or equal to 15 mm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Novilase Laser Ablation and excision (Experimental): Eligible subject will receive image-guided laser ablation of a targeted malignant breast tumor. At 4-6 weeks following the ablation, she will receive a MRI and excision. Pathology and MRI will determine rate of complete ablation. Subject is expected to proceed with radiation and/or adjuvant therapy per standard of care.
  Interventions: Device: Novilase Laser ablation

INTERVENTIONS:
Device: Novilase Laser ablation — Image-guided, percutaneous laser ablation of breast tumors

SUMMARY:
Prior to this confirmatory pivotal study, the multicenter Br-002 feasibility study was completed. 98% of tumors less than or equal to 15mm were completely ablated in one procedure.This study will evaluate Novilase for the focal destruction of malignant tumors of the breast that are less than or equal to 15 mm against a performance goal for the standard of care, lumpectomy. The ASBrS' goal of less than 20% retreatment by 2020 was selected as a representative performance goal, i.e., 80.0%, and is consistent with published effectiveness rates for lumpectomy.

DETAILED DESCRIPTION:
Subjects with biopsy-diagnosed malignant breast tumors less than or equal to 15 mm will be invited to participate. Subjects will receive a screening MRI and if eligible will then have laser ablation, followed by MRI and an excision at 4-6 weeks following the laser procedure. This study will be deemed successful if the lower limit of a 95% confidence interval for the proportion of patients who have complete tumor ablation with one Novilase laser ablation procedure at 4-6 weeks post-procedure is greater than the performance goal. Specifically, Novilase will have demonstrated success if the complete tumor ablation rate is greater than 87.85%.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 18 years and older
* Able to give written informed consent herself
* Definitive pathologic diagnosis by needle core biopsy
* Unifocal malignant tumor (T1a-c, N0-1, M0) that does not exceed 15 mm in longest dimension and measures at least 5 mm away from the skin and chest wall, or can be moved at least 5 mm away from the skin and chest wall by injection of saline or local anesthetic
* No more than 10 mm of calcifications confined to the tumor on imaging
* Tumor is well visualized through ultrasound or x-ray mammography imaging and amenable to image-guidance therapy (i.e., a tumor which is well visualized through imaging can be identified from surrounding breast tissue and does not have margins obscured by other structures or artifacts on the images)
* Tumor is well visualized on MRI
* Subject with mammographic appearance of overall dense parenchymal tissue may be included, as long as a clearly evident marker is present at tumor site
* Tumor with less than 25% intraductal component, as determined by core biopsy
* No clinically significant co-morbidities (e.g., chronic illnesses existing simultaneously with and usually independent of breast cancer) that affect life expectancy
* Subject weight limited to ≤300 lbs. or ≤136 kg
* Subject agrees to comply with standard of care radiation or adjuvant therapy as prescribed by physician

Exclusion Criteria:

* Subject younger than 18 years of age
* Pregnant or breast-feeding
* Tumor poorly visualized by ultrasound or x-ray mammography imaging
* Contraindications to administration of gadolinium-based contrast agent, including: prior allergic reaction to a gadolinium-based contrast agent, moderate to end-stage kidney disease, and/or acute or chronic severe renal insufficiency (Glomerular filtration rate (GFR) <30ml/min/1.73 sq. meters)
* Contraindications to MRI according to site guidelines (e.g., cardiac pacemaker, metallic implants)
* History of severe asthma
* Tumor measuring greater than 15 mm in longest dimension
* Microcalcifications that extend beyond target tumor such that overall longest dimension of target tumor and calcifications is longer than 15 mm.
* Advanced stage breast cancer
* Tumors that are lobular neoplasm, metastatic carcinoma to breast, sarcoma, Phyllodes tumor, or Paget's disease
* Tumor with only DCIS with microinvasion
* Extensive intraductal component in lesion (i.e., >25%) as determined by core biopsy
* Subject who is known to be BRCA positive
* Tumor that is ER/PR/HER2 negative (TNBC)
* Inability to lie in prone or supine position for one hour
* Subject who is currently participating in another investigational treatment, device or drug study through follow up that would interfere with this trial
* Subject without a definitive HER2 test according to ASCO/CAP guidelines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of target tumors completely ablated in one procedure | 4-6 weeks
  Efficacy: Rate of complete ablation by Novilase laser ablation
Frequency of adverse events (categorized using the NCI Common Terminology for Adverse Events (CTCAE) v4.0 guidelines) post-laser ablation and post-surgery | 4-6 weeks
  Safety: frequency of AEs

SECONDARY OUTCOMES:
Patient reported rate of return to activities of daily living post-laser ablation and post-surgery | 4-6 weeks
  Rate of recovery
Physician reported cosmetic satisfaction, utilizing the 4-point scoring system of breast cosmesis in protocol (e.g., excellent, good, fair, poor) post-laser ablation and post-surgery (4-6 weeks) | 4-6 weeks
  Post-procedure cosmetic satisfaction
Health related quality of life outcome measures at three timepoints via EORTC QLQ-C30 & QLQ-BR23 questionnaire (baseline and 4-6 weeks post-laser ablation and post-surgery) | 4-6 weeks
  Health-related quality of life outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: John Lewin, MD, Principal Investigator — Yale University
Locations (12):
- United States (7):
  - City of Hope, Duarte, California
  - UC San Diego Health, La Jolla, California
  - Eisenhower Health, Rancho Mirage, California
  - Yale University, New Haven, Connecticut
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Summit Health, Florham Park, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
- Germany (2):
  - St. Elisabeth-Krankenhaus Köln-Hohenlind, Cologne
  - Heidelberg University Hospital, Heidelberg
- Ichilov | Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Switzerland (2):
  - Breast Centre Zurich, Zurich
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No